CLINICAL TRIAL: NCT06414343
Title: LATe TreatmENT Related Toxicity in Melanoma (LATENT)
Acronym: LATENT
Status: Not yet recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR6009
Record Dates: First submitted 2024-04-24; First posted 2024-05-16 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational - no intervention — Observational - no intervention

SUMMARY:
Recent improvements in advanced melanoma treatment with immunotherapy have dramatically improved patient survival. Longer survival however has come at a cost of toxicity. Short term side effects can occur in >50% of patients undergoing immunotherapy treatment; however, many long-term survivors are also living with serious consequences of these treatments which may be under reported in literature.

Data regarding long term toxicities, from these treatments is lacking and an area of important unmet clinical need. Therefore, in collaboration with the Clatterbridge and Christie's teams, the investigators propose to retrospectively analyse the nature, incidence, frequency, and severity of immune related toxicities in around 400 patients who received immunotherapy for advanced melanoma with ongoing durable responses to treatment of at least 3 years.

The investigators will set up a collective anonymized database and record this information through review of electronic medical records of patients that meet the eligibility criteria. The investigators will also review the patterns of use of long-term immunosuppression and assess the need for specialist referrals for managing late side effects.

The investigators hope that this data will help us address gaps in the management of long-term survivors by identifying areas of need and establishing a coordinated evidence based multidisciplinary service to provide personalised, risk stratified long term follow up.

DETAILED DESCRIPTION:
LATENT will be a retrospective non-interventional analysis of pre-existing data from patient medical records and, therefore patients will not be required to participate in any risky procedures, treatments or hospital visits. The study will therefore not require explicit informed consent from eligible participants.

A potential ethical issue could arise around explicit consent of patients for collection and publication of their data. The investigators aim to circumvent this by only using data that has already been recorded from direct patient care.

The investigators will pseudo-anonymise personal data and mitigate risk of identification through:

1. Direct health care providers screening for eligible patients from clinic records based on clear inclusion and exclusion criteria
2. Allocation of de-identified serial numbers for patients on the database used to collect and record relevant data
3. Exportation and storage of de-identified data from all sites on a common trusted research environment (TRE) 'BRIDGE' for blinded analysis by the Research team
4. Reporting of anonymised/de-identified data only, for publication

In addition, the investigators aim to reduce selection bias by eliminating the need for explicit consent as unwell patients with greater clinical needs may be unable to consent and would not be included in the study, thereby only selecting for well patients and potentially underrepresenting a vital group of patients, compromising the scientific validity of the study.

As this is a multicentre study, de-identified, anonymised data from all centres will be exported and stored in a single secure password protected TRE for analysis. The main centre in charge of maintaining and analysing the database, with appropriate data sharing agreements with individual sites, will be The Royal Marsden team.

The investigators do not anticipate any legal issues arising from this study.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of melanoma
* Age 18 years or older
* Treated between January 2005- December 2020 with immune checkpoint inhibitor therapy including either Pembrolizumab, Nivolumab, Ipilimumab or combinations, for advanced melanoma (unresectable stage III or stage IV)
* Ongoing response to therapy of at least 3 years duration at point of study entry

Exclusion Criteria:

* Diagnoses of other concurrent malignancies needing active treatment
* Received Immune checkpoint inhibitors for non-metastatic melanoma or in the adjuvant setting only.
* Received other treatments including targeted therapy as the most recent line of treatment or following immunotherapy.
* Progression of disease on or following immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This will be a collaborative multicentre non-interventional retrospective analysis of pre-recorded data collected from patient medical records by direct treating teams. The participants will be patients of at least age 18, treated for advanced and metastatic melanoma between 2005-2020 with immune checkpoint inhibitors and have ongoing response to treatment (either stable disease, partial or complete response per RECIST 1.1) for at least 3 years at the time of inclusion in the study. Patients with metastatic melanoma treated with immunotherapy will be identified from the electronic hospital records by treating clinical teams/research team at each centre and screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To describe patterns of a range of medical late toxicities following immunotherapy treatment for advanced melanoma patients | 12 months
  • Descriptive analysis of proportion of patients (%) developing immune related adverse events in those with advanced melanoma with ongoing response of at least 3 years following treatment with immune checkpoint inhibitors. Description of severity of each type of toxicity and adverse events experienced in the overall population measured as Grade 1-5 as per Common Terminology Criteria for Adverse Events (CTCAE v5.0).

SECONDARY OUTCOMES:
Exploration of differences in proportions of patients | 12 months
  • Exploration of differences in proportions of patients developing different types and severities of late toxicities according to treatment type (single vs doublet immunotherapy), disease (stage, mutational status) and patient characteristics (eg; age, gender, smoking status, etc) using univariate and multivariate analyses.
Time to occurrence of irAEs | 12 months
  • Time to occurrence of irAEs using Kaplan-Meier survival analysis measured in years and months.
Descriptive analyses of the frequency of use of immunosuppressive agents | 12 months
  • Descriptive analyses of the frequency of use of immunosuppressive agents used (%) for treating late immune toxicities for each type of agent, toxicity and duration of immunosuppressive treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Young, MD, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, Chelsea, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No